CLINICAL TRIAL: NCT01701583
Title: Effect of Omalizumab (Xolair) on the Basophil Proteome in Patients With Chronic Idiopathic Urticaria
Brief Title: Effect of Omalizumab (Xolair) on Basophils in Patients With Chronic Idiopathic Urticaria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-0780
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Chronic Urticaria
Keywords: Chronic Idiopathic Urticaria; CIU; Urticaria; Chronic Hives; Xolair
MeSH Terms: conditions — Chronic Urticaria; Urticaria | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omalizumab (Experimental): Patients will receive omalizumab 300mg subcutaneously every 4 weeks for 12 weeks at the study center.
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — Patients will receive omalizumab 300mg subcutaneously every 4 weeks for 12 weeks at the study center.
  Other Names: Xolair

SUMMARY:
This study looks at changes in cell proteins in people with chronic hives treated with omalizumab.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate for changes in the proteins produced in white blood cells (basophils) in patients with chronic hives who are treated with and respond to omalizumab.

ELIGIBILITY:
Inclusion Criteria:

* Chronic urticaria (hives) for more than 6 weeks.
* No improvement with standard doses of antihistamines (loratadine 10 mg daily, desloratadine 5 mg daily, fexofenadine 180 mg daily, cetirizine 10 mg daily, or levocetirizine 5 mg daily)

Exclusion Criteria:

* Taken any oral steroids for 1 month prior to beginning the study.
* Taken any other immunomodulatory drugs (sulfasalazine, hydroxychloroquine, cyclosporine, methotrexate) for 1 month prior to beginning the study.
* Physical urticaria as a primary diagnosis.
* Known allergic precipitant of urticaria such as foods.
* Urticarial Vasculitis.
* Anemia.
* Asthma.
* Serum Immunoglobulin E (IgE) >700 IU/ml.
* Women of childbearing potential not using contraception method(s), as well as women who are pregnant and/or breastfeeding.
* Known sensitivity to omalizumab or this class of drug.
* Use of any other investigational agent in the last 1 month.
* Untreated intercurrent illness.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04; Primary Completion 2016-04 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Dreskin, M.D., Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Denver, Colorado, United States

REFERENCES:
- [Result] Stitt JM, Dzieciatkowska M, Edwards MG, Hansen K, Hedlund G, Dreskin SC. The basophil proteome in chronic spontaneous urticaria distinguishes responders to omalizumab from non-responders. Clin Exp Allergy. 2018 Jul;48(7):898-901. doi: 10.1111/cea.13149. Epub 2018 May 20. No abstract available. PMID 29671921

RESULTS

PARTICIPANT FLOW:
Groups:
- Omalizumab: Omalizumab 300mg subcutaneously every 4 weeks for 12 weeks
- Controls: Control subjects without urticaria who did not receive omalizumab
Period: Overall Study
Arm/Group | Omalizumab | Controls
Started | 7 | 3
Completed | 5 | 3
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline demographic data for participants who did or did not received Omalizumab are combined in order to protect the privacy of the three control participants.
Groups:
- Omalizumab: Omalizumab 300mg subcutaneously every 4 weeks for 12 weeks at the study center.
- Total: Total of all reporting groups
Arm/Group | Omalizumab | Controls | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 3 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Urticaria Activity Score for 7 days [Median (Standard Deviation); unit: units on a scale] — The Urticaria Activity Score summed over 7 days (UAS7) is a self-reported diary based measure used to assess itch severity and hive count in chronic spontaneous urticaria (CSU). Scores range from 0 to 42, with higher scores indicating more severe disease activity. Population: Only the 7 subjects with urticaria completed UAS7 scores. The 3 controls did not have urticaria.
  units on a scale
    number analyzed (Participants) | 7 | 0 | 7
    (all) | 30 (11) |  | 30 (11)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Basophil Proteome
Description: In patients with chronic urticaria who respond clinically to omalizumab, the proteome of blood basophils will be measured at baseline (pre-treatment) and at weeks 6 and 13 (post-treatment). The number of participants with a change observed in basophil proteome out of the total number of participants, stratified by responders and non-responders, is reported.
Time Frame: Baseline through week 13
Population: There were 7 subjects with chronic urticaria treated with omalizumab and 3 control subjects without chronic urticaria, not treated with omalizumab. There was insufficient data for weeks 6 and 13 to analyze primary outcome.
Measure: Count of Participants; unit: Participants
Groups:
- Omalizumab Responders: Subjects with chronic urticaria, treated with omalizumab who responded to the drug
- Controls: Subjects without chronic urticaria, not treated with omalizumab
- Omalizumab Non-responders: Subjects with chronic urticaria, treated with omalizumab who did not respond to the drug
Arm/Group | Omalizumab Responders | Controls | Omalizumab Non-responders
Number analyzed (Participants) | 4 | 3 | 3
Participants
  Baseline | 4 | 0 | 3
  Week 6: number analyzed (Participants) | 0 | 0 | 0
  Week 13: number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change in Basophil Proteome in Responders to Omalizumab Compared to Non-responders to Omalizumab.
Description: Change in basophil proteome in responders to omalizumab compared to non-responders to omalizumab. However, there was insufficient data from weeks 6 and 13 to analyze this outcome.
Time Frame: Baseline through week 13
Population: There were 7 subjects with chronic urticaria treated with omalizumab and 3 control subjects without chronic urticaria, not treated with omalizumab. Because the data from subsequent time points was not able to be analyzed, the investigators were unable to analyze this outcome because no change comparison could be made.
Arm/Group | Omalizumab Responders | Controls
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to week 13
Arm/Group | Omalizumab | Controls
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 3/7 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omalizumab (N=7) | Controls (N=3)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Flushing (Endocrine disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Unable to assess primary or secondary outcome due to insufficient data at weeks 6 and 13.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No